CLINICAL TRIAL: NCT04812821
Title: Statement of Care of Anemia in Delivering Patients at Nord Franche-Comte Hospital
Acronym: ANEMIA
Status: Completed | Type: Observational
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-02
Record Dates: First submitted 2021-03-16; First posted 2021-03-24 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2021-03

CONDITIONS: Pregnancy Anemia
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — questionnaire post delivery

SUMMARY:
Anemia is a common pregnancy condition that has multiple origins. Its frequency and severity seem to be increasing, despite the existing management recommendations and the awareness of health professionals. The objective of this study is to make a statement of this pathology within our establishment, to evaluate the proportion of patients presenting this pathology and to highlight possible risk factors.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Delivery at Nord Franche-Comte Hospital
* Delivery ≥ 32 weeks of amenorrhea
* Informed patient and non-opposition of participation

Exclusion Criteria:

* Protected adults (Patients under guardianship, curatorship, safeguard of justice or under family authorization)
* Medical interruption of pregnancy
* Patients with fetal death in utero or neonatal death
* Minor patients
* Premature delivery before 32 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presenting eligibility criteria and giving birth at NFC Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1177 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Estimation of the proportion of patients presenting anemia during delivery | 6 month
  Percentage of patients with hemoglobin less than 10.5 g/dl at entry into the delivery room

SECONDARY OUTCOMES:
Risk factors underlying anemia during delivery with a large questionnaire | 6 month
  Link between presence or absence of anemia and type of follow-up (gynecological or midwife, anemia during pregnancy and iron supplementation strategy and compliance), living conditions (geographical origin, socioeconomic situation, diet) and comorbidities

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Nord Franche-Comté, Trévenans, France

IPD SHARING:
Plan to Share IPD: No